CLINICAL TRIAL: NCT07280065
Title: Diagnostic Testing of Post-Traumatic Stress Disorder (PTSD) Using the Senseye Diagnostic Tool in Adults : United States, Australia, and Decentralized Trial (DCT) Protocol
Brief Title: REVEAL Study - Diagnostic Testing for PTSD Using the Senseye Diagnostic Tool
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Senseye, Inc. (Industry)
Collaborators: Lindus Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CSP-002
Record Dates: First submitted 2025-11-21; First posted 2025-12-12 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: PTSD - Post Traumatic Stress Disorder
Keywords: PTSD; Trauma; MDD; Depression; GAD; Anxiety; Nightmares; Major Depressive Disorder; Avoidance
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic; Wounds and Injuries; Depression; Anxiety Disorders; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Participants will be evaluated for PTSD presence and severity using both the CAPS-5-R structured clinical interview [the clinical reference standard] and the Senseye Diagnostic Tool (DT) [the study device]. The order of these interventions will be randomized - some participants will be assessed with the CAPS-5-R first and Senseye DT second, while others will be assessed with the Senseye DT first and CAPS-5-R second.
Masking Description: It is not possible to mask the intervention being given to participants. However, during the pivotal (test validation) phase of the study, investigators and the sponsor will be masked/blinded to the intervention output (PTSD results). Participants will always be masked/blinded to the intervention output.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- PTSD assessment comparing the Senseye DT to the clinical reference standard (Experimental): All participants enrolled will be administered both the Senseye DT and the CAPS-5-R. The CAPS-5-R is used as the study's clinical reference standard to establish the "ground truth" for PTSD presence and severity. The order of administration will be randomized.
  Interventions: Device: Senseye Diagnostic Tool (DT); Behavioral: Clinician Administered PTSD Scale for DSM-5, Revised Version

INTERVENTIONS:
Device: Senseye Diagnostic Tool (DT) — Software as a Medical Device - the Senseye DT is an investigational diagnostic device that is an application which can be installed on iPhones 13 and newer. The device administers various tasks on the phone screen that the participant completes while video and/or audio is recorded (depending on the task). Recordings are analyzed by a machine learning algorithm to predict the presence and severity of PTSD.
Behavioral: Clinician Administered PTSD Scale for DSM-5, Revised Version — The CAPS-5-R is a standardized stuctured clinical interview for determining PTSD presence and severity. It is a behavioral interview administered by a trained mental health clinician or clinical rater. Participant responses to various questions about traumatic experiences and resulting symptoms are scored to determine PTSD presence according to DSM-5 criteria and PTSD severity according to the CAPS-5-R severity scale.
  Other Names: CAPS-5-R

SUMMARY:
The goal of the REVEAL PTSD study is to test how well the Senseye DT works as a diagnostic test for Post-traumatic Stress Disorder (PTSD) in adults 18 and older who are experiencing one or more symptoms that might be related to PTSD.

The Senseye DT is software as a medical device (SaMD) and is an iPhone app that administers a series of simple tasks on the phone while recording video during the tasks through the front-facing camera. The videos are analyzed by a a Machine Learning (ML) algorithm to identify physiologic signals that might be indicative of PTSD. Data collected in this study will be used to train and tune the ML algorithm, then test it for accuracy.

The main questions this study aims to answer are:

1. How accurate is the Senseye DT in detecting PTSD compared to structured clinical interviews, the current clinical standard for diagnostic testing?
2. How accurately does the Senseye DT predict PTSD severity?
3. How fast is the Senseye DT to use compared to structured clinical interviews?

Participants will attend a virtual screening visit via video call to determine eligibility and consent to participate. Once enrolled, participants will attend 2 or 3 additional study visits:

* Visit 1: A virtual visit where standard mental health assessments will be given by clinical raters trained in mental health and administering these structured clinical interviews. These assessments include the Structured Interview Guide for the Montgomery-Asburg Depression Rating Scale (SIGMA), the Structured Interview Guide for the Hamilton Anxiety Scale (SIGH-A), and the MINI International Neurodiagnostic Interview. The Clinician-Administered PTSD Scale for DSM-5 Revised Version (CAPS-5-R) may also be conducted, if randomly selected.
* Visit 2: A visit to use the Senseye DT. For participants near one of the study's physical site locations, this visit will be done in person at the site. For all others, this visit will be conducted virtually.
* Visit 3: For participants not randomly selected to have the CAPS-5-R administered at Visit 1, a third and final visit will be scheduled for this assessment. This visit will be conducted virtually.

The total expected participation time for enrolled participants is 6-7 hours over the course of 2-3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is willing and able to read, understand, and sign the approved Informed Consent Form (ICF).
2. Age 18 years old or older.
3. In the past month, participant presents with at least one of the following:

   * nightmares or unwanted, intrusive thoughts
   * avoidance of specific thoughts or situations
   * feelings of being constantly on guard, watchful, or easily startled
   * feeling numb or detached from people, activities, or surroundings; and/or
   * persistent feelings of guilt or self blame for things that have happened.
   * excessive anxiety and worry (apprehensive expectation), occurring more days than not for at least 6 months, about a number of events or activities (such as work or school performance)
   * sleep disturbance (difficulty falling or staying asleep, or restless unsatisfying sleep)
   * depressed mood: most of the day, nearly every day, feeling sad, empty, or hopeless
   * markedly diminished interest or pleasure in activities: loss of interest or pleasure in most activities, nearly every day
   * self-report of significant weight loss or gain and/or changes in appetite
   * insomnia or hypersomnia: sleeping too little or too much
   * psychomotor agitation or retardation: observable restlessness or slowed movements
   * abnormal fatigue or loss of energy: feeling tired or lacking energy more than usual
4. Deemed likely to comply with the study protocol by the study team, including willing communication of adverse events (AEs), mental health history, current and past psychiatric medication & treatments, and ability to attend all study visits.
5. Participant agrees to provide emergency contact information at Screening Visit and their physical location at each visit (if they are joining the visit remotely).
6. Participant is psychologically stable as determined by the investigator or delegate.
7. Participant has access to the following:

   * a device with stable internet and Wi-Fi connection capable of supporting video calls (e.g., tablet, computer with webcam, etc.)
   * a second smart device that must be an iPhone 13 or newer (Not inclusive of the iPhone13 Mini)
8. Participant home/environment meets criteria for Senseye DT setup (remote visits only)

Exclusion Criteria:

1. Current diagnosis of epilepsy and/or other seizure disorders.
2. A history of at Screening OR positive at Visit 1 for bipolar I or II, mania, or one or more schizophrenia-spectrum or other psychotic disorders, including schizophrenia, schizoaffective disorder, delusional disorder, psychotic depression, and psychosis.
3. Compromised facial neuro-ophthalmic integrity (e.g., due to stroke, MS, ALS, or other neurological conditions).
4. Current diagnosis of dementia, delirium, amnestic disorders, autism, hydrocephalus, posterior cortical atrophy, aphasia, multiple sclerosis, or stroke-related cognitive dysfunction.
5. Current eye disorders which prevent the patient from using the Senseye DT:

   * Vision impairment preventing ability to read with correction (including corneal disease, dense cataract, diabetic retinopathy, macular degeneration, glaucoma, etc.).
   * Use of corrective lenses including glasses and contacts is permitted. Colored contacts and cosmetic lenses that obscure or enhance the pupil are not permitted.
   * Significant eye lid droop blocking the pupil.
   * Persistent blurry vision, headaches, and/or light sensitivity resulting from conditions including abnormal pupil dilation or reactivity (e.g, mydriasis).
   * Recent eye surgeries (within 2 weeks) or planned eye surgeries within the study duration.
   * Intraocular inflammation, including iritis and anterior uveitis.
   * Ocular trauma resulting in uncorrected or permanent bilateral damage.
6. Active suicidal and/or homicidal intent or other self-injurious behavior which may put the participant and/or others at risk per the investigator's clinical judgement, or has suicidal ideation of level 4 or 5 as determined by the C-SSRS.
7. Suicidal behavior within the last year as determined by the C-SSRS at the time of screening.
8. Significant suicidal ideation within the last 6 months as determined by ideation of level 4 or 5 by the C-SSRS at the time of screening.
9. Current reported usage (within 2 weeks of Screening Visit and/or planned ongoing usage during the study) of psychotropic drugs and/or non-psychotropic drugs or medication which may affect use of the Senseye DT:

   * Narcotics/opioids (e.g., Heroin, Vicodin, oxycodone, codeine, Tramadol, etc.).
   * Tricyclic antidepressants (TCAs) (e.g., Tofranil, Pamelor, amitriptyline, doxeprin, etc.).
   * Monoamine Oxidase Inhibitors (MAOIs) (e.g., Emsam, Parnate, Nardil, Marplan, etc.).
   * Select antihypertensive medications (alpha-2 receptor agonists, clonidine, peripheral adrenergic inhibitors, Alpha & Beta blockers, and Rauwolfia alkaloids). Note: If Prazosin can be abstained from for > 24 hours prior to the Senseye DT visit, the exclusion does not apply for that medication.

   Stimulants (e.g., Amphetamines, Ritalin, Focalin, pseudoephedrine/Sudafed, ecstasy, cocaine, methamphetamines, cathinones, etc.). Note: Caffeine or nicotine use is not exclusionary. Note: that if Sudafed, pseudoephedrine, and stimulants commonly used to treat ADHD (e.g., Ritalin, Focalin, Adderall, etc. can be abstained from for > 24 hours prior to the Senseye DT visit, the exclusion does not apply for those medications.
   * Psychedelics/psychotomimetics (Lysergic acid, psilocybin, mescaline, phencyclidine, methoxetamine, etc.).
   * Cholinergic or anticholinergic agents (e.g., Urecholine, Pilocar, Aricept, Miostat, Evoxac, ipratropium/Atrovent, oxybutynin/Ditropan, scopolamine, etc.), except antihistamines other than Benadryl or diphenhydramine. Note: If Benadryl/diphenhydramine can be abstained from for > 24 hours prior to the Senseye DT visit, the exclusion does not apply.
   * Spravato or Ketamine.
   * Eye drops unless the participant is able to abstain from use for > 72 hours prior to the Senseye DT visit. Note: Artificial tears can be used if needed during the Senseye DT use.
   * Central Nervous System (CNS) depressants (Benzodiazepines and Barbiturates)
10. Current reported usage (within 2 weeks of Screening Visit and/or planned ongoing usage during the study) of vagal nerve stimulation, deep brain stimulation, transcranial magnetic stimulation, or other stimulation or energy-based therapies.
11. Any condition which precludes the ability for patients to safely and accurately complete clinical assessments, questionnaires, or to follow instructions necessary to administer the Senseye DT (e.g., significant developmental disabilities, language disorders, cognitive deficiencies, or other neurodevelopmental disorders).
12. Medical diagnosis of Traumatic Brain Injury (TBI) within the last 12 months based on participant self-report.
13. Lifetime history of any of the following: surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system (CNS) disorder (e.g., Alzheimer's Disease, Parkinson's Disease), or any other disease/procedure/accident/intervention that, according to the clinician, is deemed associated with significant injury to, or malfunction of, the CNS.
14. Involved in active litigation related to the participant's psychiatric symptoms
15. Pregnancy as determined by self-report.
16. Currently incarcerated.
17. Participant requires a legal authorized representative to consent.
18. Prior enrollment in this study or in other Senseye Machine Learning (ML) studies within the last 12 months.
19. Unwilling or unable to comply with all study related procedures, in the opinion of the investigator, including medical and non-medical procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1900 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the Senseye DT as an objective PTSD diagnostic test | Baseline
  Performance goals (lower bound of 95% confidence intervals) are set to ≥0.70 sensitivity and ≥0.70 specificity for the device's binary PTSD diagnostic test result as compared to the Clinical Reference Standard. The Senseye DT would provide a clear, objective diagnostic result that is 70% of the research-quality structured clinical interview accuracy (70% of 100% accuracy). This level of accuracy is clinically sufficient for providing a meaningful diagnostic output for PTSD as it provides an accuracy equivalent to current standard-of-care methods in mental healthcare. In primary care settings where a majority of PTSD patients are initially seen for symptoms, the Senseye DT would provide a 50% improvement in accuracy compared to current methods (70% vs. 20%).

SECONDARY OUTCOMES:
Time to administer the Senseye DT compared to the clinical reference standard | Baseline
  Intended to demonstrate a statistically significant difference in time to administer the Senseye DT compared to the CAPS-5-R structured clinical interview. It is expected that the Senseye DT time to administer will be ~73% faster (24 min. vs. 90 min.) compared to the CAPS-5-R. This time difference represents a clinical benefit compared to existing methods, as a research-quality assessment for PTSD with accuracy equivalent to current real-world standard of care can be delivered in less time.
Agreement between the Senseye DT PTSD severity score output and the CAPS-5-R severity scale | Baseline
  Intended to validate the Senseye DT's capability to output a PTSD severity rating. A valid output will be a Senseye DT severity output that is shown to be correlated with the CAPS-5-R severity rating via a regression analysis.
Sensitivity and specificity of the Senseye DT used as an objective test for PTSD symptoms that would benefit from evidence-based treatment. | Baseline
  Endpoint is intended to compare the Senseye DT binary output (PTSD-positive, PTSD-negative) to the presence of clinically-relevant severity based on the CAPS-5-R severity outcome. A CAPS-5-R cutoff score will be established to define clinically-relevant severity (i.e., symptom severity necessitating treatment). This endpoint differs from the Primary Endpoint as the Primary Endpoint is based on the presence of DSM-5-defined PTSD while this endpoint is based on the presence of a symptom severity necessitating treatment (regardless of the presence of DSM-5 PTSD).

OTHER OUTCOMES:
Number of Serious Adverse Device Effects (SADEs). | Baseline to study completion, an average of 2 weeks.
  Evaluate the number of SADEs occurring during the trial related or possibly related to the Senseye DT.
Device positive predictive value (PPV) and negative predictive value (NPV). | Baseline
  Evaluate the PPV and NPV for the Senseye DT.
Participant satisfaction for using the Senseye DT compared to the CAPS-5-R structured clinical interview. | Baseline
  Evaluate participant preference information and satisfaction for using the Senseye DT compared to the CAPS-5-R. Data will be collected on participant-completed surveys.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Savannah VA Clinic, Savannah, Georgia
  - Velocity Clinical Research, Meridian, Idaho
  - Lowcountry Center for Veterans Research, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No